CLINICAL TRIAL: NCT02470936
Title: A Randomized Clinical Trial of Web-based Lifestyle Tools and Resources Versus Usual Care Among Men With Prostate Cancer
Brief Title: Web-based Lifestyle Trial Among Men With Prostate Cancer: Prostate 8
Acronym: Prostate 8
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: American Cancer Society, Inc. (Other); Prostate Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-13555
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1- Lifestyle Intervention (Experimental): Men will receive a web-based, personalized lifestyle program. They will receive personalized prostate cancer-specific lifestyle recommendations on specific habits based on their eligibility survey responses. They will have access to the website composed of four topic areas (get active, eat well, stop smoking, and find support), receive a Fitbit and access to a Fitbit account and community group, and receive text messages and refrigerator magnet to reinforce behaviors. The website will be updated frequently with new tips and material and two weekly blogs will be maintained. Final content is reviewed by study investigators and patient advocates. Men will complete an intervention acceptability survey (acceptability of the website and intervention components) at 3 months.
  Interventions: Behavioral: Lifestyle intervention
- Group 2 - Control (No Intervention): Men randomized to the control group will receive standard of care. They will receive access to the website and personalized lifestyle recommendations on the 8 healthy habits targeted in the study after the 3 month trial.

INTERVENTIONS:
Behavioral: Lifestyle intervention — Patients will have access to the lifestyle website and an activity monitor (e.g., Fitbit), receive texts, and be provided with individualized lifestyle recommendations.
  Arms: Group 1- Lifestyle Intervention

SUMMARY:
A randomized controlled trial of a technology-based lifestyle intervention vs. usual care among men with low-risk prostate cancer to determine the feasibility and acceptability of the intervention and the effect of the intervention on behavior change related to exercise, diet, and not smoking.

DETAILED DESCRIPTION:
This is a PI-initiated, randomized, unblinded, clinical trial of a technology-based 3 month lifestyle intervention vs. usual care among men with low risk prostate cancer. We will recruit and consent 76 men with prostate cancer at UCSF. The subjects will be asked to complete questionnaires, 7 days accelerometer measurement, body measurements (weight, waist, hip, pulse, blood pressure) and collection of blood specimen at baseline and 3 months. Subjects will be randomized into two arms (Intervention Group and Control Group). The Intervention Group (N=38) will have access to the lifestyle website and an activity monitor (e.g., Fitbit), receive text messages, and be provided with individualized lifestyle recommendations. The Control Group (N=38) will have standard of care and be asked to continue with their usual lifestyle habits. They will receive access to the lifestyle website and be provided with individualized lifestyle recommendations at 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. clinical stage ≤T3a nonmetastatic prostate cancer within 5 years
2. completion of treatment ≥3 months prior to enrollment, if not on active surveillance
3. ability to walk unassisted
4. be able to speak and read English
5. ability to navigate websites and email, and have internet access
6. able to travel to UCSF for pre- and post-study blood collection

Exclusion Criteria:

1. any contraindications to moderate or vigorous aerobic exercise
2. psychiatric condition preventing the patient from giving informed consent or adhering to the study protocol
3. reporting adherence to more than 4 of the 8 targeted lifestyle behaviors via questionnaires at screening

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Fitbit use | 3 months
  We will measure the number of days the Fitbit was used during the study period in the intervention arm only to assess study feasibility
text message use | 3 months
  We will measure the number of text messages responded to that required a reply in the intervention arm only during the study period to assess study feasibility
website use - number of days the website was visited | 3 months
  We will measure the total number of days the website was visited in the intervention arm only during the study period to assess study feasibility
website use - number of website visits | 3 months
  We will measure the total number of website visits in the intervention arm only during the study period to assess study feasibility
intervention acceptability | 3 months
  We will assess intervention acceptability via questionnaire at 3 months in the intervention group.
self-reported change in health behaviors | 3 months
  We will assess change in health behaviors via questionnaire at baseline and 3 months.

SECONDARY OUTCOMES:
change in physical activity measured by activity monitor | 3 months
  This is assessed via 7-day accelerometer measurements at baseline and 3 months.
change in task self-efficacy | 3 months
  We will assess confidence in performing behaviors via questionnaire at baseline and 3 months.
change in plasma antioxidant Vitamin E | 3 months
  We will assess Vitamin E levels at baseline and 3 months.
change in plasma antioxidant lycopene | 3 months
  We will assess lycopene levels at baseline and 3 months.
change in fasting glucose | 3 months
  We will assess fasting glucose at baseline and 3 months.
change in cholesterol | 3 months
  We will assess cholesterol at baseline and 3 months.
change in hemoglobin A1c | 3 months
  We will assess hemoglobin A1c at baseline and 3 months.
change in C-reactive protein | 3 months
  We will assess C-reactive protein at baseline and 3 months.
change in waist circumference | 3 months
  We will assess waist circumference at baseline and 3 months.
change in weight | 3 months
  We will assess weight at baseline and 3 months.
change in body mass index | 3 months
  We will assess body mass index at baseline and 3 months.
depression | 3 months
  Center for Epidemiologic Studies Depression Scale completed at baseline and 3 months.
anxiety | 3 months
  Memorial Anxiety Scale for Prostate Cancer and State Anxiety completed at baseline and 3 months. Trait anxiety completed at baseline.
health-related quality of life | 3 months
  Expanded Prostate Cancer Index Composite-26 and Short Form Health Survey-36 completed at baseline and 3 months.
maintenance or adoption of self-reported behaviors after 1 year | 1 year
  We will assess change in health behaviors via questionnaire at baseline, 3 months, and 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Kenfield, ScD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco (UCSF), San Francisco, California, United States

REFERENCES:
- [Background] Kenfield SA, Van Blarigan EL, Ameli N, Lavaki E, Cedars B, Paciorek AT, Monroy C, Tantum LK, Newton RU, Signorell C, Suh JH, Zhang L, Cooperberg MR, Carroll PR, Chan JM. Feasibility, Acceptability, and Behavioral Outcomes from a Technology-enhanced Behavioral Change Intervention (Prostate 8): A Pilot Randomized Controlled Trial in Men with Prostate Cancer. Eur Urol. 2019 Jun;75(6):950-958. doi: 10.1016/j.eururo.2018.12.040. Epub 2019 Jan 10. PMID 30638635